CLINICAL TRIAL: NCT03003884
Title: A Study of Remimazolam Tosilate in Patients Undergoing Diagnostic Upper GI Endoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HR-RMZL-IIc-UGE
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2016-12

CONDITIONS: Sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- Remimazolam Tosilate 1 (Experimental): IV of Remimazolam Tosilate at 5mg for initial dose
  Interventions: Drug: Remimazolam Tosilate
- Remimazolam Tosilate 2 (Experimental): IV of Remimazolam Tosilate at 7mg for initial dose
  Interventions: Drug: Remimazolam Tosilate
- Remimazolam Tosilate 3 (Experimental): IV of Remimazolam Tosilate at 8mg for initial dose
  Interventions: Drug: Remimazolam Tosilate
- Remimazolam Tosilate 4 (Experimental): IV of Remimazolam Tosilate at 5mg for initial dose.At the end of the endoscopy, flumazenil was injected.
  Interventions: Drug: Remimazolam Tosilate
- Propofol (Active Comparator): IV of Propofol at 1.5mg/kg for initial dose
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam Tosilate — Initial dose plus supplemental doses as necessary.
  Arms: Remimazolam Tosilate 1; Remimazolam Tosilate 2; Remimazolam Tosilate 3; Remimazolam Tosilate 4
Drug: Propofol — Initial dose plus supplemental doses as necessary.
  Arms: Propofol

SUMMARY:
The purpose of this study is to find out the optimal dose for Remimazolam Tosilate as a procedural sedative during a diagnostic upper GI endoscopy and to assess its efficacy and safety profile comparing to propofol.

DETAILED DESCRIPTION:
This is an multi-center,single-blinded,parallel-group,dose-finding study using Remimazolam or propofol for sedation in patients undergoing diagnostic upper GI endoscopy.Subjects are randomized to different treatment groups (including 4 for Remimazolam Tosilate and 1 for propofol).Lidocaine and fentanyl are permitted during a diagnostic upper GI endoscopy.Efficacy and safety profiles of Remimazolam Tosilate are to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 18-60 years；
* intending to undergo diagnostic upper GI endoscopy
* American Society of Anesthesiologists Physical Status Score (ASA PS) I or II；
* 18 kg/m²<BMI(Body Mass Index)<30 kg/m².

Exclusion Criteria:

* Patients with a suspected upper GI bleed an conditions predisposing to hemorrhage at the discretion of the investigator;
* one or more of the laboratory findings fall out of the limitations for this study(platelet,hemoglobin,aspartate aminotransferase,etc.);
* history of recent use of narcotics,analgesics,anaesthetics and benzodiazepine hypnotics;
* history of severe cardiovascular disease;
* cerebral disease or mental disorder;
* allergic to drugs used in the study;
* pregnant women or those in lactation period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
successful sedation rate as measured by the proportion of subjects who experienced successful sedation during diagnostic upper GI endoscopy. | From start of study drug injection to patient discharge (approx. 3 hours)

SECONDARY OUTCOMES:
recovery time as measured by time | After the last of study drug injection to patient discharge (approx. 3 hours)
rate of hypotension as measured by the proportion of subjects who experienced hypotension during a diagnostic upper GI endoscopy | From start of study drug injection to patient discharge (approx. 3 hours)
rate of hypoxaemia as measured by the proportion of subjects who experienced hypoxaemia during a diagnostic upper GI endoscopy | From start of study drug injection to patient discharge (approx. 3 hours)
rate of respiratory depression as measured by the proportion of subjects who experienced respiratory depression during a diagnostic upper GI endoscopy | From start of study drug injection to patient discharge (approx. 3 hours)
pain on injection was assessed by the patient immediately after administration of the study drug | 1-10 minutes (from the beginning of sedation )]

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Union Medical College Hospital, Beijing, Beijing Municipality, China